CLINICAL TRIAL: NCT02617680
Title: Factors Affecting the Effective End-tidal Concentration of Desflurane Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, Principal Investigator, University Hospital Hradec Kralove
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201404515P
Record Dates: First submitted 2015-11-15; First posted 2015-12-01 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: General Anesthetic Drug Adverse Reaction
Keywords: Desflurane; end tidal concentration; age; anesthesia
MeSH Terms: interventions — Air; Desflurane; Nitric Oxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- desflurane - oxygen in air (Experimental): The manufacturer recommended age-corrected end-tidal concentrations of desflurane in air should be set and achieved initially. Concentration of oxygen should be 50%.
  Interventions: Drug: desflurane - oxygen in air
- desflurane - oxygen in nitric oxide (Experimental): The manufacturer recommended age-corrected end-tidal concentrations of desflurane with nitric oxide - oxygen should be set and achieved initially.Concentration of oxygen should be 50%.
  Interventions: Drug: desflurane - oxygen in nitric oxide

INTERVENTIONS:
Drug: desflurane - oxygen in air — The manufacturer recommended age-corrected end-tidal concentrations of desflurane in air should be set and achieved initially. Individual EEtC of desflurane will be defined according to entropy parameters and maintained in the targeted range of static and response entropy 40-50
  Other Names: suprane
  Arms: desflurane - oxygen in air
Drug: desflurane - oxygen in nitric oxide — The manufacturer recommended age-corrected end-tidal concentrations of desflurane with nitric oxide - oxygen should be set and achieved initially. Individual EEtC of desflurane will be defined according to entropy parameters and maintained in the targeted range of static and response entropy 40-50
  Other Names: suprane
  Arms: desflurane - oxygen in nitric oxide

SUMMARY:
There is accumulating evidence that inappropriate depth of anaesthesia is associated with increased risk of postoperative complications including risk of death. The aim of this study was to identify factors determining the effective end-tidal concentration (EEtC) of desflurane, duration of wash in and wash out phase, and to estimate the risk of perioperative awareness in patients undergoing elective neurosurgical procedure.

DETAILED DESCRIPTION:
All patients with American Society of Anesthesiologists (ASA) physical status I-III scheduled for elective neurosurgical procedure under general anaesthesia are studied. In each individual, the manufacturer recommended age-corrected end-tidal concentrations of desflurane is set and achieved initially. Individual effective end-tidal concentration (EEtC) of desflurane is then defined according to entropy parameters and maintained in the targeted range of static and response entropy 40-50. Effective analgesia is maintained according to surgical plethysmographic index (SPI) and dose of muscle relaxants according to neuromuscular transmission monitoring (TOF). Comorbidity, regular intake of alcohol and medication, smoking, sex, weight, height, and age are recorded. Postoperative questionnaire is used to reveal the intraoperative awareness.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* elective neurosurgical procedure under general anaesthesia
* Age between 18 and 78
* elective procedures with estimated duration 1 - 3 hours

Exclusion Criteria:

* Glasgow coma scale GCS below 14
* other rhythm than sinus
* pacemaker stimulation
* planned postoperative ventilation

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
end tidal concentration of desflurane according to age | from the start of procedure up to 4 hours

SECONDARY OUTCOMES:
Time to spontaneous ventilation | from end of anesthesia up to 1 hour
Time to extubation | from the end of anesthesia up to 1 hour
Time to reaction to command | from the end of anesthesia up to 1 hour
Wash in phase | up to achievement of manufacturer age-corrected end-tidal concentrations of desflurane up to 10 minutes
  sec
Wash out phase | from the end of procedure up to 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Vlasta Dostalova, MD., Ph.D., Principal Investigator — University Hospital Hradec Kralove, Czech Republic
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia